CLINICAL TRIAL: NCT04910165
Title: Adductor Canal Blocks Using Exparel for Pain Control After Total Knee Arthroplasty
Brief Title: Exparel Use in Adductor Canal Block After Total Knee Arthroplasty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Luke's Hospital, Pennsylvania (Other)
Responsible Party: Principal Investigator, Chinenye Nwachuku, Principal Investigator, St. Luke's Hospital, Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SLIR 2019-106
Record Dates: First submitted 2021-05-25; First posted 2021-06-02 (Actual); Results first posted 2022-05-20 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Arthritis Knee; Pain, Postoperative; Opioid Use
Keywords: Exparel; adductor; knee; arthroplasty; opioid
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Exparel (Experimental): Liposomal Bupivacaine use as active ingredient in the block
  Interventions: Drug: Exparel
- Control (Active Comparator): Ropivacaine use as active ingredient in the block
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Exparel — Exparel used in Adductor Canal Block plus Infiltration Between Popliteal Artery and Capsule of Knee using Ropivacaine
  Arms: Exparel
Drug: Ropivacaine — Ropivacaine used in Adductor Canal Block plus Infiltration Between Popliteal Artery and Capsule of Knee using Ropivacaine
  Arms: Control

SUMMARY:
Exparel has been shown to have better pain control compared to previously used infiltration agents, including bupivacaine, while having a minor side effect profile. The purpose of this study is to explore the effectiveness of Exparel (liposomal bupivacaine) in Adductor Canal Blocks for peri-operative pain control following a total knee arthroplasty (TKA) procedure.

DETAILED DESCRIPTION:
The effectiveness of an Exparel Block (Bupivacaine Liposomal Injectable Suspension) for post-operative pain control has been well studied with encouraging results. At the investigators' institution, Exparel has been approved as a safe and effective option for use in shoulder surgeries and have had encouraging results in adductor canal use for pain control in patients undergoing TKA. Exparel has been shown to have better pain control compared to previously used infiltration agents, including bupivacaine, while having a minor side effect profile. The purpose of this study is to explore the effectiveness of Exparel (liposomal bupivacaine) in Adductor Canal Blocks (ACB) for peri-operative pain control following a total knee arthroplasty (TKA) procedure. Specifically, the investigators look to see if Exparel ACB reduces opioid requirement use post-operatively, reduces pain scores post-operatively, provides earlier mobilization, and decreases length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients were eligible for inclusion if they were undergoing unilateral primary TKA for a diagnosis of knee osteoarthritis and were not undergoing any additional concomitant procedures were.

Exclusion Criteria:

* Patients were not eligible for our study if they were undergoing revision TKA, if they were undergoing bilateral TKA or concomitant procedures, or if they had an active infection.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chinenye Nwachuku, MD, Principal Investigator — St. Luke's Hospital and Health Network, Pennsylvania
Locations (1):
- St. Luke's University Health Network, Bethlehem, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients that presented to our outpatient Orthopaedic clinic and signed up to undergo a Total Knee Arthroplasty (TKA) were eligible for our study. No additional advertising was used.
Period: Overall Study
Arm/Group | Exparel | Control
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exparel | Control | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Full Range); unit: years] | 66.1 [46 to 80] | 66.2 [43 to 83] | 66.2 [43 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 29 | 54
  Male | 25 | 21 | 46
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100
BMI [Mean (Full Range); unit: kg/m^2] | 32.2 [20.98 to 41.89] | 32.3 [23.89 to 44.02] | 32.25 [20.98 to 44.02]
American Society of Anesthesiology (ASA) Score [Count of Participants; unit: Participants] — Determined by hospital Anesthesia team based on guidelines set forward by the American Society of Anesthesiologists ASA 1: A normal healthy patient. ASA 2: A patient with mild systemic disease. ASA 3: A patient with severe systemic disease. ASA 4: A patient with severe systemic disease that is a constant threat to life.
  ASA 5: A moribund patient who is not expected to survive without the operation. NOTE: Higher numbers are worse grades
  Participants
    ASA 2 | 26 | 26 | 52
    ASA 3 | 24 | 24 | 48
Smoking [Count of Participants; unit: Participants]
  Yes | 10 | 9 | 19
  No | 40 | 41 | 81
Kellgren and Lawrence Osteoarthritis Grade [Count of Participants; unit: Participants] — K&L 0: No radiographic findings of osteoarthritis K&L 1: Doubtful narrowing of joint space and possible osteophytic lipping K&L 2: Definite osteophytes and possible narrowing of joint space K&L 3: Moderate multiple osteophytes, definite narrowing of joint space, small pseudocystic areas with sclerotic walls and possible deformity of bone contour K&L 4: Large osteophytes, marked narrowing of joint space, severe sclerosis, and definite deformity of bone contour.
  NOTE: Higher grades denote more advanced arthritis.
  Participants
    2 | 5 | 9 | 14
    3 | 29 | 24 | 53
    4 | 16 | 17 | 33
Previous Surgery [Count of Participants; unit: Participants]
  Yes | 16 | 11 | 27
  No | 34 | 39 | 73
Previous TKA [Count of Participants; unit: Participants]
  Yes | 10 | 9 | 19
  No | 40 | 41 | 81

OUTCOME MEASURES:

1. Primary Outcome: Hospital Length of Stay
Description: Inpatient post-operative stay after undergoing TKA procedure
Time Frame: Through entire inpatient hospital stay (lasted from 1 day to 1 week)
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Exparel | Control
Number analyzed (Participants) | 50 | 50
Hours | 36.3 (12.4) | 49.7 (35.3)
Statistical Analysis 1: Comparison: Exparel vs Control; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney) — p-values reported are calculated by the listed statistical test

2. Primary Outcome: Inpatient Opioid Use
Description: Opioid usage during their inpatient post-operative hospital stay
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: Milimorphine Equivalents/Day
Arm/Group | Exparel | Control
Number analyzed (Participants) | 50 | 50
Milimorphine Equivalents/Day | 40.9 (20.7) | 47.3 (27.9)
Statistical Analysis 1: Comparison: Exparel vs Control; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney) — p-values reported are calculated by the listed statistical test

3. Primary Outcome: Numeric Rating Scale (NRS) Pain Score Improvement
Description: Measured with Numerical Rating Scale (Range: 0-10, Minimum:0, Maximum:10). Change in NRS Pain Score from pre-operative levels. Positive changes indicate a decrease in pain levels from pre-operative levels.
Time Frame: 6 weeks
Population: Number of patients available in Post-operative day (POD) 2 lower secondary to earlier discharges. Number of patients available for analysis in in POD 7-42 time points secondary to their follow up). To account for this, both an "intention to treat" and a "per protocol" analysis were completed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exparel | Control
Number analyzed (Participants) | 50 | 50
units on a scale
  POD 0 | 1.8 (2.7) | -0.2 (2.7)
  POD 1 | 1.0 (2.7) | -1.3 (2.4)
  POD 2: number analyzed (Participants) | 12 | 27
  POD 2 | 2.3 (2.6) | -0.1 (2.3)
  POD 7: number analyzed (Participants) | 44 | 44
  POD 7 | 1.8 (3.5) | 0.2 (2.9)
  POD 14: number analyzed (Participants) | 38 | 40
  POD 14 | 3.2 (3.2) | 1.3 (3.0)
  POD 28: number analyzed (Participants) | 37 | 38
  POD 28 | 3.9 (2.6) | 2.2 (2.9)
  POD 42: number analyzed (Participants) | 36 | 38
  POD 42 | 5.2 (2.7) | 3.0 (2.5)
Statistical Analysis 1: Comparison: Exparel vs Control; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney) — p-values reported are calculated by the listed statistical test

4. Primary Outcome: Outpatient Opioid Use
Description: Opioid usage in the immediate post-operative period after hospital discharge
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Milimorphine Equivalents/Day
Arm/Group | Exparel | Control
Number analyzed (Participants) | 50 | 50
Milimorphine Equivalents/Day | 33.4 (11.6) | 32.1 (13.2)
Statistical Analysis 1: Comparison: Exparel vs Control; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney) — p-values reported are calculated by the listed statistical test

5. Primary Outcome: WOMAC Score
Description: Western Ontario and McMaster Universities Osteoarthritis Index Patient Subjective Outcome Score (Range: 0-96, Minimum:0, Maximum:96). Subsections include Pain (Range:0-20, Minimum:0, Maximum:20), Stiffness (Range:0-8; Minimum:0, Maximum:8), and Functional Limitation (Range0-68, Minimum:0, Maximum:68). Measured as change in score from baseline levels. Positive scores indicate an improvement in WOMAC scores from pre-operative levels.
Time Frame: 6 weeks
Population: Number of patients available for analysis in in POD 7-42 time points decreased secondary to their follow up. To account for this, both an "intention to treat" and a "per protocol" analysis were completed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exparel | Control
Number analyzed (Participants) | 44 | 44
units on a scale
  POD 7 Pain Subscore | 4.0 (4.8) | 1.2 (5.7)
  POD 7 Stiffness Subscore | 1.5 (2.7) | 0.2 (2.8)
  POD 7 Physical Function Subscore | 14.8 (19.0) | 4.6 (17.3)
  POD 7 Total Score | 20.3 (24.8) | 6.0 (23.6)
  POD 14 Pain Subscore: number analyzed (Participants) | 38 | 40
  POD 14 Pain Subscore | 6.2 (5.0) | 4.2 (5.4)
  POD 14 Stiffness Subscore: number analyzed (Participants) | 38 | 40
  POD 14 Stiffness Subscore | 2.2 (2.3) | 0.7 (2.8)
  POD 14 Physical Function Subscore: number analyzed (Participants) | 38 | 40
  POD 14 Physical Function Subscore | 22.6 (13.6) | 14.7 (17.6)
  POD 14 Total Score: number analyzed (Participants) | 38 | 40
  POD 14 Total Score | 31.1 (19.4) | 19.6 (24.2)
  POD 28 Pain Subscore: number analyzed (Participants) | 37 | 38
  POD 28 Pain Subscore | 7.2 (4.5) | 6.7 (4.3)
  POD 28 Stiffness Subscore: number analyzed (Participants) | 37 | 38
  POD 28 Stiffness Subscore | 2.5 (2.6) | 1.7 (2.5)
  POD 28 Physical Function Subscore: number analyzed (Participants) | 37 | 38
  POD 28 Physical Function Subscore | 26.2 (14.1) | 21.2 (14.9)
  POD 28 Total Score: number analyzed (Participants) | 37 | 38
  POD 28 Total Score | 36.0 (19.3) | 29.7 (20.2)
  POD 42 Pain Subscore: number analyzed (Participants) | 37 | 38
  POD 42 Pain Subscore | 9.8 (4.2) | 7.4 (5.0)
  POD 42 Stiffness Subscore: number analyzed (Participants) | 37 | 38
  POD 42 Stiffness Subscore | 4.2 (1.9) | 2.8 (2.1)
  POD 42 Physical Function Subscore: number analyzed (Participants) | 37 | 38
  POD 42 Physical Function Subscore | 34.1 (11.8) | 25.5 (11.6)
  POD 42 Total Score: number analyzed (Participants) | 37 | 38
  POD 42 Total Score | 48.2 (16.4) | 35.7 (17.1)
Statistical Analysis 1: Comparison: Exparel vs Control; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney) — p-values reported are calculated by the listed statistical test

6. Secondary Outcome: Number of Participants Needing to be Readmitted to the Hospital Secondary to Inadequate Pain Control Post-operatively
Description: Rate of needing to be readmitted to the hospital secondary to inadequate pain control post-operatively at any point during the study period.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Exparel | Control
Number analyzed (Participants) | 50 | 50
Participants | 2 | 6
Statistical Analysis 1: Comparison: Exparel vs Control; Test type: Superiority; p < 0.05, Fisher Exact — p-values reported are calculated by the listed statistical test

7. Secondary Outcome: Number of Participants Needing to be Admitted to an Inpatient Rehabilitation Facility Post-Operatively
Description: Rate of needing to be discharged to an inpatient rehabilitation facility after TKA procedure secondary to inadequate pain control and functional recovery
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Exparel | Control
Number analyzed (Participants) | 50 | 50
Participants | 3 | 4
Statistical Analysis 1: Comparison: Exparel vs Control; Test type: Superiority; p < 0.05, Fisher Exact — p-values reported are calculated by the listed statistical test

ADVERSE EVENTS:
Time Frame: 17 months (June 2020-October 2021) Each patient was assessed for adverse events by direct history and physical exam by investigators at POD 0, POD 1, POD 2, POD 7, POD 14, POD 28, and POD 42.
Description: Clinicaltrials.gov definitions will be used
Arm/Group | Exparel | Control
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 4/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exparel (N=50) | Control (N=50)
Nausea and Vomiting (General disorders) | 0 (0) | 4 (4)

LIMITATIONS AND CAVEATS:
Block efficacy is dependent on the performing anesthesiologist, with multiple performing anesthesiologists introducing variability that was not accounted for. The use of drains was surgeon specific rather than part of our study protocol. The state's online drug monitoring program reports narcotic prescriptions filled but not necessarily taken possibly pointing to a discrepancy. Finally, all patients were obtained from one demographic area, and all surgeries were only performed by two surgeons

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/65/NCT04910165/Prot_SAP_001.pdf